CLINICAL TRIAL: NCT00000648
Title: A Pilot Study Evaluating Penicillin G and Ceftriaxone as Therapies for Presumed Neurosyphilis in HIV Seropositive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 145
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Neurosyphilis
Keywords: Penicillin G; Neurosyphilis; Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Ceftriaxone
MeSH Terms: conditions — HIV Infections; Neurosyphilis; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Penicillin G; Ceftriaxone

INTERVENTIONS:
Drug: Penicillin G potassium
Drug: Ceftriaxone sodium

SUMMARY:
To provide information on the response of HIV infected, neurosyphilis patients to the currently recommended treatment for neurosyphilis; to determine whether possible co-infection with both HIV and syphilis makes more difficult the diagnosis of syphilis; to explore the usefulness of an alternative treatment which, if effective, would permit outpatient treatment for neurosyphilis that until now required prolonged hospitalization.

Studies suggest that syphilis treatment failures may be more common in HIV infected patients than in patients without HIV infection and that treatment failures occur due to and/or are displayed as central nervous system (CNS) involvement. Very little is known about the best treatment course for neurosyphilis in patients who are also infected with HIV.

DETAILED DESCRIPTION:
Studies suggest that syphilis treatment failures may be more common in HIV infected patients than in patients without HIV infection and that treatment failures occur due to and/or are displayed as central nervous system (CNS) involvement. Very little is known about the best treatment course for neurosyphilis in patients who are also infected with HIV.

HIV infected patients who are presumed to have neurosyphilis or have definitive neurosyphilis are treated for the neurosyphilis with either penicillin G or ceftriaxone. Patients are treated for 10 days and followed for 50 weeks after treatment. Patients receiving penicillin G are hospitalized while receiving the penicillin. Patients receiving ceftriaxone are treated on an inpatient basis for at least the first three days and may then be discharged to receive outpatient treatment. During treatment, patients are permitted to take antiretroviral drugs or other drugs for opportunistic infections except for drugs that are antisyphilitic. Lumbar punctures will be performed.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral drugs.
* Concurrent treatment for opportunistic infections with non-antisyphilitic drugs.
* Metronidazole, aminoglycosides, trimethoprim / sulfamethoxazole (TMP / SMX), polymyxin, vancomycin, dapsone, pentamidine, acyclovir, antifungals, clindamycin, immunomodulators, and quinolones.

Patients must:

* Have HIV infection.
* Have presumable or documented neurosyphilis.
* Be capable of giving informed consent.
* Have life expectancy of at least 52 weeks.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* History of penicillin or cephalosporin immediate hypersensitivity reaction characterized by angioneurotic edema, hyperemia, urticaria, bronchospasm, and/or anaphylaxis.
* History of mucosal or blistering rash in response to related treatment.

Concurrent Medication:

Excluded:

* Antitreponemal therapy (amoxicillin, doxycycline, tetracycline hydrochloride, erythromycin, procaine penicillin, any beta lactam, or chloramphenicol).

Patients with the following are excluded:

* Other etiology of cerebrospinal (CSF) abnormalities other than HIV and syphilis infection in patients who present with clinical symptoms (this is not required in asymptomatic patients).

Prior Medication:

Excluded:

* Treatment for syphilis within 1 year prior to study entry.
* Antitreponemal therapy (amoxicillin, doxycycline, tetracycline hydrochloride, erythromycin, procaine penicillin, any beta lactam, or chloramphenicol) within 45 days prior to study entry.

Unwilling or unable to comply with follow-up schedule, including repeat lumbar punctures.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Study Completion 1996-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hook EW III, Study Chair
Locations (42):
- United States (42):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Yale Univ / New Haven, New Haven, Connecticut
  - Florida Keys Memorial Hosp, Key West, Florida
  - Med Service, Miami, Florida
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Robert Wood Johnson Med School/UMDNJ, New Brunswick, New Jersey
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Nassau County Med Ctr, East Meadow, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Montefiore Drug Treatment Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Family Health Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Samaritan Village Inc / Bronx Municipal Hosp, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - North Central Bronx Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Wake Med Ctr / Univ of North Carolina, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Med Univ of South Carolina / UNC, Charleston, South Carolina
  - Northwest Family Ctr at the Harbor View Med Ctr, Seattle, Washington
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Silva MG, Cruz ML, Lopes GB, Leite CG, Menezes JA. Neurosyphilis in HIV patients. Int Conf AIDS. 1996 Jul 7-12;11(2):280 (abstract no ThB4170)